CLINICAL TRIAL: NCT05634889
Title: The T-REX-Trial: Tailored Regional External Beam Radiotherapy in Clinically Node-negative Breast Cancer Patients With 1-2 Sentinel Node Macrometastases; an Open, Multicenter, Randomized Non-inferiority Phase 3-trial.
Brief Title: The T-REX Trial: Tailored Regional External Beam Radiotherapy in Clinically Node-negative Breast Cancer Patients With 1-2 Sentinel Node Macrometastases.
Acronym: T-REX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-05093-02
Record Dates: First submitted 2022-11-18; First posted 2022-12-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; radiotherapy; gene expression analysis; adjuvant breast cancer treatment; regional breast cancer treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Radiotherapy to the remaining breast after breast conserving surgery or chest wall after mastectomy, and regional axillary lymph node levels I-IV. Internal mammary nodes are included in the target volume if the tumor has a central/medial localization in the breast.
- Intervention (Experimental): No regional radiotherapy. Radiotherapy is given to the remaining breast after breast conserving surgery. Chest wall radiotherapy after mastectomy only in case of wide spread multifocality.
  Interventions: Radiation: De-escalation

INTERVENTIONS:
Radiation: De-escalation — No regional radiotherapy. Radiotherapy is given to the remaining breast after breast conserving surgery. Chest wall radiotherapy after mastectomy only in case of wide spread multifocality.
  Arms: Intervention

SUMMARY:
T-REX is a randomized multicenter, non-inferiority trial.

Aim: To evaluate whether regional radiotherapy may safely be omitted in clinically node negative breast cancer patients with one or two sentinel node macrometastases and an estrogen receptor positive, HER2-negative tumor. Leading to an improved quality of life and reduced side effects, without worsening recurrence free survival at five years.

Intervention: Patients will be randomized to locoregional radiotherapy towards the breast/chestwall and regional lymph nodes vs. to a de-escalated radiotherapy.

In the intervention arm no lymph node irradiation will be given. Radiotherapy is still given to the remaining breast after breast conserving surgery, but no radiotherapy is given after mastectomy.

Sample size: 1350 patients

Primary end-point: Recurrence free survival at five years.

Gene expression analysis: For all patients gene expression analysis for the gene signatures ARTIC, POLAR and OncotypeDX will be performed and related to risk of recurrence and benefit of adjuvant radiotherapy.

DETAILED DESCRIPTION:
In this multicenter, prospective randomized trial clinically node-negative breast cancer patients with 1-2 macrometastases in their sentinel lymph node biopsy, and an estrogen receptor positive, HER2-negative tumor, will be randomly assigned to either receive adjuvant locoregional radiotherapy, or no regional radiotherapy.

The main aim is to evaluate whether regional radiotherapy may safely be omitted in patients with limited lymph node metastasis and an estimated low risk of locoregional recurrence. Recurrence free survival after five years is the primary outcome, which for non-inferiority should not worsen more than 4.5 percentage units. Secondary outcomes are locoregional recurrence, regional nodal recurrence, new contralateral BC, distant recurrence free survival, overall survival, non-breast malignancies, cardiac disease, arm morbidity, and health-related quality of life.

Target volumes include:

Standard arm - The remaining breast/chest wall, axillary lymph node levels I-III, the supraclavicular lymph nodes (level IV), the interpectoral lymph nodes and in patients with a medial/central tumor also the internal mammary lymph nodes.

Intervention arm - The remaining breast after breast conserving surgery. No radiotherapy after mastectomy

ELIGIBILITY:
Inclusion Criteria:

1. Primary unifocal or multifocal invasive breast cancer T1-T2.
2. Clinically N0.
3. Macrometastasis (>2mm) in 1-2 lymph nodes at sentinel node biopsy.
4. Oral and written consent.
5. Age ≥ 18 years.
6. All resection margins are tumor free (no tumor on ink).
7. Primary tumor ER-positive, HER2-negative.

Exclusion Criteria:

1. Regional or distant metastases outside the ipsilateral axilla.
2. Previous RT towards the planned target area, i.e. the ipsilateral chest/lymph nodes.
3. Neoadjuvant systemic therapy.
4. Axillary lymph node dissection or other previous axillary surgery on the affected side.
5. Prior history of invasive breast cancer.
6. Pregnancy.
7. Bilateral invasive breast cancer.
8. Contraindication for radiotherapy or systemic treatment.
9. Inability to absorb or understand the contents of the informed consent form; for example, through disability, inadequate language skills or dementia.
10. Other invasive cancer within 5 years prior to breast cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | Five years

SECONDARY OUTCOMES:
Locoregional recurrence | Five years
Regional nodal recurrence | Five years
New contralateral breast cancer | Five years
Distant recurrence free survival | Five years
Overall survival | Five years
Arm morbidity | Five years
  Assessed by questionnaires completed by study participants digitally or on paper between randomization and start of RT, and after 1, 3, and 5 years. The questionnaire used is the Lymphedema Functioning, Disability and Health Questionnaire (Lymph-ICF) developed by Devoogdt in 2011.
Health-related quality of life | Five years
  Assessed by the questionnaire EORTC QLQ-C-30 completed by study participants between randomization and RT, and after 1, 3, and 5 years.
Health-related quality of life | Five years
  Assessed by the questionnaire BR-23 completed by study participants between randomization and RT, and after 1, 3, and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Alkner, Associate professor, Principal Investigator — Lunds Universitet
Locations (26):
- Norway (9):
  - Ålesund, Ålesund
  - Bergen, Bergen
  - Bodø, Bodø
  - Gjövik, Gjøvik
  - Kristiansand, Kristiansand
  - Oslo, Oslo
  - Stavanger, Stavanger
  - Tromsø, Tromsø
  - Trondheim, Trondheim
- Sweden (17):
  - Region Västragötaland, Borås
  - Region Gävleborg, Gävle
  - Region Västra Götaland, Gothenburg
  - Region Halland, Halmstad
  - Region Jönköping, Jönköping
  - Region Kalmar län, Kalmar
  - Region Värmland, Karlstad
  - Region Östergötland, Linköping
  - Region Skåne, Lund
  - Region Örebro, Örebro
  - Region Västragötaland, Skövde
  - Region Stockholm, Stockholm
  - Region Västernorrland, Sundsvall
  - Region Västerbotten, Umeå
  - Region Uppsala, Uppsala
  - Region Kronoberg, Vaxjo
  - Region Västmanland, Västerås

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request by the T-REX study group through primary investigator Sara Alkner (sara.alkner@med.lu.se) as specified below.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The above information is available. IPD will be shared upon reasonable request after publication of the main endpoint. No end date.
Access Criteria: Study protocol, Statistical Analysis Plan, Informed Consent Form and Clinical Study Report will be available to all interested.
  Deidentified participant data, and access to biological material, could be made available to researchers who provide a methodologically sound proposal with all prepared documents for ethical approval to the T-REX study group / the T-REX biobank group through primary investigator Sara Alkner (sara.alkner@med.lu.se).

REFERENCES:
- [Derived] Alkner S, de Boniface J, Lundstedt D, Mjaaland I, Ryden L, Vikstrom J, Bendahl PO, Holmberg E, Sackey H, Wieslander E, Karlsson P. Protocol for the T-REX-trial: tailored regional external beam radiotherapy in clinically node-negative breast cancer patients with 1-2 sentinel node macrometastases - an open, multicentre, randomised non-inferiority phase 3 trial. BMJ Open. 2023 Sep 26;13(9):e075543. doi: 10.1136/bmjopen-2023-075543. PMID 37751948